CLINICAL TRIAL: NCT01739517
Title: Efficacy and Safety of Omega-3 Lipid Therapy in Pediatric Patients With Parenteral Nutrition-Associated Liver Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amarnath, Rathna, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND104555
Record Dates: First submitted 2012-11-28; First posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Short Bowel Syndrome; Cholestasis
Keywords: Short bowel syndrome; Cholestasis; Omegaven; Parenteral nutrition-associated Liver Disease
MeSH Terms: conditions — Short Bowel Syndrome; Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven Therapy (Experimental): After baseline labs, which have been collected no earlier than seven days prior to the initiation of therapy are obtained, therapy with Omegaven will be initiated at a starting dose of 0.5 g/kg/day infused over 12 hours. If tolerated, the dose will be increased to 1 g/kg/day, the goal dose. Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition.
  Interventions: Drug: Omegaven Therapy

INTERVENTIONS:
Drug: Omegaven Therapy — After baseline labs, which have been collected no earlier than seven days prior to the initiation of therapy are obtained, therapy with Omegaven will be initiated at a starting dose of 0.5 g/kg/day infused over 12 hours. If tolerated, the dose will be increased to 1 g/kg/day, the goal dose. Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition.

SUMMARY:
This pilot study seeks to demonstrate the efficacy of an intravenous lipid preparation high in omega-3 fatty acids (Omegaven) in the treatment of cholestasis in parenteral nutrition dependent patients with short gut syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be dependent upon parenteral nutrition (PN)
* Patient will have short gut syndrome (loss of >50% of small bowel)
* Patient's guardian/caregiver provides informed consent for patient to receive therapy
* Pediatric patient ≤ 1 year of age
* Expected PN duration is greater than 30 days
* Direct bilirubin >2.0 mg/dL measured on two occasions no more than one week apart

Exclusion Criteria:

* Liver dysfunction secondary to cause other than PN verified by standard of care diagnostic procedures and lab work to rule out alternative causes of neonatal cholestasis.
* Any patient in whom Omegaven therapy would be contraindicated, such as an allergy to any seafood product, egg protein, and/or previously established allergy to Omegaven
* impaired lipid metabolism
* severe hemorrhagic disorder
* unstable diabetes mellitus
* collapse and shock, stroke/embolism, recent cardiac infarction, or undefined coma status

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver dysfunction as measured by time to achieve 50 % decrease in direct bilirubin | weekly then biweekly data collection
  Direct bilirubin will be collected at baseline, then weekly for 30 days, and then biweekly, thereafter, up to an expected average of 108 weeks

SECONDARY OUTCOMES:
a) Maintenance of nutritional status | Labwork will be collected at baseline, then weekly for the first month. Thereafter, a lipid panel will be collected every 2 months, complete metabolic panel every 2 weeks, and essential fatty acid profile monthly, up to an expected average of 108 weeks
  Nutritional status will be monitored by reviewing complete metabolic panel, magnesium, weight, vitals, phosphorus, prealbumin, lipid panel, and essential free fatty acid profile. The essential fatty acid profile will be checked at baseline and then monthly for at least 6 months until the patient is determined to be receiving at least 2.7% of caloric intake from linoleic acid. If the patient's essential fatty acid profile indicates that the patient is absorbing adequate amounts of essential fatty acid, the essential fatty acid profile will be discontinued .
Occurrence of potential adverse side effects | biweekly labwork up to an expected average of 108 weeks
  Adverse events may include but are not limited to prolonged prothrombin time, hypertriglyceridemia, and anaphylaxis in relation to the patient's therapy.
c) Resolution of liver dysfunction | weekly complete metabolic panel for the first month and then biweekly thereafter, up to an expected average of 108 weeks
  Resolution of liver dysfunction will be defined by achievement of normal direct bilirubin, aspartate aminotransferase and alanine transaminase.

CONTACTS AND LOCATIONS:
Overall Officials: Terra R Varner, PharmD, Principal Investigator — Palmetto Health Children's Hospital
Locations (1):
- Palmetto Health Children's Hospital, Columbia, South Carolina, United States

REFERENCES:
- [Background] Christensen RD, Henry E, Wiedmeier SE, Burnett J, Lambert DK. Identifying patients, on the first day of life, at high-risk of developing parenteral nutrition-associated liver disease. J Perinatol. 2007 May;27(5):284-90. doi: 10.1038/sj.jp.7211686. Epub 2007 Mar 8. PMID 17344923
- [Background] Diamond IR, Sterescu A, Pencharz PB, Wales PW. The rationale for the use of parenteral omega-3 lipids in children with short bowel syndrome and liver disease. Pediatr Surg Int. 2008 Jul;24(7):773-8. doi: 10.1007/s00383-008-2174-0. Epub 2008 May 27. PMID 18504595
- [Background] Kelly DA. Intestinal failure-associated liver disease: what do we know today? Gastroenterology. 2006 Feb;130(2 Suppl 1):S70-7. doi: 10.1053/j.gastro.2005.10.066. PMID 16473076
- [Background] Gura KM, Duggan CP, Collier SB, Jennings RW, Folkman J, Bistrian BR, Puder M. Reversal of parenteral nutrition-associated liver disease in two infants with short bowel syndrome using parenteral fish oil: implications for future management. Pediatrics. 2006 Jul;118(1):e197-201. doi: 10.1542/peds.2005-2662. PMID 16818533
- [Background] Moss RL, Das JB, Ansari G, Raffensperger JG. Hepatobiliary dysfunction during total parenteral nutrition is caused by infusate, not the route of administration. J Pediatr Surg. 1993 Mar;28(3):391-6; discussion 396-7. doi: 10.1016/0022-3468(93)90238-g. PMID 8468653
- [Background] Chen WJ, Yeh SL, Huang PC. Effects of fat emulsions with different fatty acid composition on plasma and hepatic lipids in rats receiving total parenteral nutrition. Clin Nutr. 1996 Feb;15(1):24-8. doi: 10.1016/s0261-5614(96)80257-3. PMID 16843991
- [Background] de Meijer VE, Le HD, Meisel JA, Gura KM, Puder M. Parenteral fish oil as monotherapy prevents essential fatty acid deficiency in parenteral nutrition-dependent patients. J Pediatr Gastroenterol Nutr. 2010 Feb;50(2):212-8. doi: 10.1097/MPG.0b013e3181bbf51e. PMID 20038849
- [Background] Colomb V, Jobert-Giraud A, Lacaille F, Goulet O, Fournet JC, Ricour C. Role of lipid emulsions in cholestasis associated with long-term parenteral nutrition in children. JPEN J Parenter Enteral Nutr. 2000 Nov-Dec;24(6):345-50. doi: 10.1177/0148607100024006345. PMID 11071594
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of fish oil and safflower oil emulsions on diet-induced hepatic steatosis in rats receiving total parenteral nutrition. Clin Nutr. 1996 Apr;15(2):80-3. doi: 10.1016/s0261-5614(96)80024-0. PMID 16844003
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Puder M, Valim C, Meisel JA, Le HD, de Meijer VE, Robinson EM, Zhou J, Duggan C, Gura KM. Parenteral fish oil improves outcomes in patients with parenteral nutrition-associated liver injury. Ann Surg. 2009 Sep;250(3):395-402. doi: 10.1097/SLA.0b013e3181b36657. PMID 19661785